CLINICAL TRIAL: NCT00737009
Title: An Observational Study of Adherence to Adjuvant Anastrozole Therapy in Postmenopausal Patients With Early Breast Cancer Over One Year Follow-up.
Brief Title: An Observational Study of Adherence to Anastrozole in Early Breast Cancer Treatment
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Luu, Thi Khanh Trang, Study Leader, AstraZeneca Pharmaceuticals
Other Study IDs: NIS-OVN-ARI-2008/1
Record Dates: First submitted 2008-08-15; First posted 2008-08-18 (Estimated); Last update posted 2011-06-22 (Estimated); Status verified 2011-06

CONDITIONS: Breast Cancer
Keywords: Breast cancer; adherence; anastrozole; post-menopausal women
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The purpose of this study is to describe adherence to anastrozole treatment current practice: cases where anastrozole treatment was halted ( timescale and causes) and estimate the proportion of postmenopausal women with early breast cancer who continue anastrozole therapy after one year follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal woman with early breast cancer who are prescribed with anastrozole as adjuvant endocrine therapy under the routine clinical practice.
* Histologically or cytologically proven to be HR+(ER or PR +)
* No other concomitant endocrine therapy such as estrogen therapy or selective estrogen receptor modulators
* Provision of written informed consent

Exclusion Criteria:

* Recurrence of breast cancer
* Known hypersensitivity to anastrozole or to any of its excipients
* Any severe concomitant condition which makes it undesirable for the patient to participate in the trial or which would jeopardize adherence with the trial protocol: Amenorrhea<12 months and a intact uterus; Previous inclusion in the present study; Participation in a other clinical study during the last 30 days·
* Women who does not agreed to participate the program

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The target study population comprised of postmenopausal women with early breast cancer who were treated with anastrozole for at least one month and are willing to give written informed consent to participate.
Sampling Method: Probability Sample
Enrollment: 259 (Actual)
Dates: Start 2008-08; Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
To describe adherence to anastrozole treatment current practice: cases where anastrozole treatment was halted ( timescale and causes) | every 3- 6 months (4 visit in one year)

SECONDARY OUTCOMES:
Estimate the proportion of postmenopausal women with early breast cancer who continue anastrozole therapy after one year follow-up | every 3- 6 months (4 visit in one year)
Identify predictors of non- adherence | every 3- 6 months (4 visit in one year)
The proportion of DFS after 1 year follow-up | every 3- 6 months (4 visit in one year)
Describe menopausal symptoms | every 3- 6 months (4 visit in one year)

CONTACTS AND LOCATIONS:
Overall Officials: Nguyen Van Dinh, MD, Principal Investigator — K Hospital Hanoi, Vietnam; Tran Nguyen Ha, Principal Investigator — HCMC Cancer Hospital; Tran Dang Khoa, Principal Investigator — Hanoi Cancer Hospital; Ton That Cau, Principal Investigator — Hue Central Hospital
Locations (3):
- Vietnam (3):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City
  - Research Site, Huế